CLINICAL TRIAL: NCT00161551
Title: A Randomized, Prospective Multicenter Study to Determine the Incidence of Atrial Fibrillation and Heart Failure in Correlation to Stimulation Modes of Pacemakers
Brief Title: Mode Evaluation in Sick Sinus Syndrome Trial (MODEST)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medtronic BRC (Industry)
Collaborators: Vitatron GmbH (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MODEST V.2.2.1
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2011-08-02 (Estimated); Status verified 2006-10

CONDITIONS: Sick Sinus Syndrome
Keywords: Cardiac Pacing, artificial; Atrial Fibrillation; Heart Failure; Pacemaker leads; Pacing Mode
MeSH Terms: conditions — Sick Sinus Syndrome; Atrial Fibrillation; Heart Failure

INTERVENTIONS:
Device: Vitatron T70 DR

SUMMARY:
The purpose of this study is to determine the incidence of atrial fibrillation and heart failure in patients with pacemaker therapy with different pacing modes (AAI, DDD, and a novel algorithm to minimize ventricular pacing).

DETAILED DESCRIPTION:
Background: Dual-chamber pacemaker therapy has become the mainstay for treating symptomatic sick sinus syndrome (SSS). This approach aims to results in a physiologic conduction pattern, while protecting against atrioventricular conduction anomalies. Smaller studies and subgroup analyses of larger trials suggest that ventricular stimulation associated with this treatment has adverse effects, especially an increased incidence of atrial fibrillation and heart failure.

Methods: In MODEST, a study on patients with sick sinus syndrome who have an indication for pacing therapy, atrial pacing (AAI) is compared with dual-chamber pacing (DDD) combined with a novel algorithm developed to lower the number of ventricularly paced beats. The study aims to assess the impact of ventricular pacing on the development of atrial arrhythmias and to test the hypothesis that DDD pacing using the algorithm is associated with a higher rate of atrial arrhythmias as atrial pacing. Included will be patients with SSS and no high degree AV node disease except for patients with first-degree AV block ≤300ms. Patients will be followed stratified by their Wenckebach point (≥ 120 bpm versus < 120 bpm).

Conclusion: MODEST is a large, prospective, randomized, multicenter trial aiming to compare a novel type of dual-chamber pacing approach (that includes an algorithm designed to lower the number of ventricularly paced beats) with pure atrial pacing, assessing the impact on the incidence of atrial arrhythmias in patients with sick sinus syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic sinus bradycardia, Sinusarrest
* Symptomatic SA block
* Bradycardia-Tachycardia-Syndrome
* Binodal diseases

Exclusion Criteria:

* 1st degree AV Block
* 2nd degree AV block
* 3rd degree AV block
* Total right bundle branch block
* Indication for biventricular stimulation
* Inter atrial conduction delays (P-wave > 150MS)
* Permanent or therapy refractory Atrial Fibrillation
* Heart Failure acc. NYHA III or IV
* Myocardial Infarction less than 6 months before pacemaker implant
* Hypertrophic obstructive cardiomyopathy
* Symptomatic hypo- or hyperthyreosis
* Cardiogenic shock
* Pregnancy
* Lactation period
* Unstable angina pectoris
* Poorly controlled Diabetes mellitus
* Neuromuscular diseases
* Patients under 18 years of age
* Patients involved in other studies
* Reduced expectancy of life due to other diseases
* Patients who cannot attend follow-up visits regularly

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Estimated)
Dates: Start 2004-11; Study Completion 2010-12

PRIMARY OUTCOMES:
Primary objective is to assess how the pacing mode affects the incidence of atrial fibrillation (AF) in patients with sick sinus syndrome. Since there are no data on the safety of AAI pacing in patients with Wenckebach points < 120 bpm and accor

SECONDARY OUTCOMES:
Number of patients with atrial fibrillation or heart failure > NYHA II
AF burden
Symptomatic atrial fibrillation
Time period to first recurrence of AF
Number of patients without recurrence of AF
Mean duration of sinus rhythm
Course of Wenckebach point
Second- and third-degree AV block
Reprogramming from AAI to DDD
Fraction of atrial versus ventricular pacing
Safety of treatment, complications
Number of cardioversions
Patients with persistent atrial fibrillation (AF >48h)
Patients with permanent atrial fibrillation (AF throughout the follow-up period)
Hospital admissions for cardiac reasons

CONTACTS AND LOCATIONS:
Overall Officials: Volker Schibgilla, MD, Principal Investigator
Locations (5):
- Germany (5):
  - Klinikum Coburg, Coburg
  - Universitätskrankenhaus Eppendorf, Hamburg
  - Kardiologische Gemeinschaftspraxis, Papenburg
  - Kardiologische Praxis, Starnberg-Percha
  - Sophien- und Hufelandklinikum GmbH, Weimar

REFERENCES:
- [Background] Lamas GA, Orav EJ, Stambler BS, Ellenbogen KA, Sgarbossa EB, Huang SK, Marinchak RA, Estes NA 3rd, Mitchell GF, Lieberman EH, Mangione CM, Goldman L. Quality of life and clinical outcomes in elderly patients treated with ventricular pacing as compared with dual-chamber pacing. Pacemaker Selection in the Elderly Investigators. N Engl J Med. 1998 Apr 16;338(16):1097-104. doi: 10.1056/NEJM199804163381602. PMID 9545357
- [Background] Lamas GA, Lee KL, Sweeney MO, Silverman R, Leon A, Yee R, Marinchak RA, Flaker G, Schron E, Orav EJ, Hellkamp AS, Greer S, McAnulty J, Ellenbogen K, Ehlert F, Freedman RA, Estes NA 3rd, Greenspon A, Goldman L; Mode Selection Trial in Sinus-Node Dysfunction. Ventricular pacing or dual-chamber pacing for sinus-node dysfunction. N Engl J Med. 2002 Jun 13;346(24):1854-62. doi: 10.1056/NEJMoa013040. PMID 12063369
- [Background] Andersen HR, Nielsen JC, Thomsen PE, Thuesen L, Mortensen PT, Vesterlund T, Pedersen AK. Long-term follow-up of patients from a randomised trial of atrial versus ventricular pacing for sick-sinus syndrome. Lancet. 1997 Oct 25;350(9086):1210-6. doi: 10.1016/S0140-6736(97)03425-9. PMID 9652562
- [Background] Nielsen JC, Kristensen L, Andersen HR, Mortensen PT, Pedersen OL, Pedersen AK. A randomized comparison of atrial and dual-chamber pacing in 177 consecutive patients with sick sinus syndrome: echocardiographic and clinical outcome. J Am Coll Cardiol. 2003 Aug 20;42(4):614-23. doi: 10.1016/s0735-1097(03)00757-5. PMID 12932590
- [Background] Connolly SJ, Kerr CR, Gent M, Roberts RS, Yusuf S, Gillis AM, Sami MH, Talajic M, Tang AS, Klein GJ, Lau C, Newman DM. Effects of physiologic pacing versus ventricular pacing on the risk of stroke and death due to cardiovascular causes. Canadian Trial of Physiologic Pacing Investigators. N Engl J Med. 2000 May 11;342(19):1385-91. doi: 10.1056/NEJM200005113421902. PMID 10805823
- [Background] Mattioli AV, Vivoli D, Mattioli G. Influence of pacing modalities on the incidence of atrial fibrillation in patients without prior atrial fibrillation. A prospective study. Eur Heart J. 1998 Feb;19(2):282-6. doi: 10.1053/euhj.1997.0616. PMID 9519322
- [Background] Kerr CR, Connolly SJ, Abdollah H, Roberts RS, Gent M, Yusuf S, Gillis AM, Tang AS, Talajic M, Klein GJ, Newman DM. Canadian Trial of Physiological Pacing: Effects of physiological pacing during long-term follow-up. Circulation. 2004 Jan 27;109(3):357-62. doi: 10.1161/01.CIR.0000109490.72104.EE. Epub 2004 Jan 5. PMID 14707022
- [Background] Wilkoff BL, Cook JR, Epstein AE, Greene HL, Hallstrom AP, Hsia H, Kutalek SP, Sharma A; Dual Chamber and VVI Implantable Defibrillator Trial Investigators. Dual-chamber pacing or ventricular backup pacing in patients with an implantable defibrillator: the Dual Chamber and VVI Implantable Defibrillator (DAVID) Trial. JAMA. 2002 Dec 25;288(24):3115-23. doi: 10.1001/jama.288.24.3115. PMID 12495391